CLINICAL TRIAL: NCT06534853
Title: Comparison of Post Facilitation Stretch Versus Reciprocal Inhibition in Quadratus Lumborum Syndrome: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/22
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Quadratus Lumborum Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFS Group (Experimental): Group A along with Post facilitation stretch of quadratus lumborum will a comprehensive therapeutic regimen that includes a 10-minute session of hot pack therapy specifically targeted at the low back region. In addition to this, participants will receive trigger point release therapy to alleviate muscle tension. The treatment plan also incorporates a tailored exercise protocol designed to enhance back health and strength. This protocol includes:
  1. Back isometric exercises
  2. Bridging exercises
  3. Cat and camel stretches
  4. Prone press-ups
  5. Abductor strengthening exercises
  Interventions: Other: Post Facilitation Stretch; Other: Conventional Physical Therapy
- RI Group (Experimental): Group B along with Reciprocal inhibition of quadratus lumborum will a comprehensive therapeutic regimen that includes a 10-minute session of hot pack therapy specifically targeted at the low back region. In addition to this, participants will receive trigger point release therapy to alleviate muscle tension. The treatment plan also incorporates a tailored exercise protocol designed to enhance back health and strength. This protocol includes:
  1. Back isometric exercises
  2. Bridging exercises
  3. Cat and camel stretches
  4. Prone press-ups
  5. Abductor strengthening exercises
  Interventions: Other: Reciprocal Inhibition; Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Post Facilitation Stretch — The patient is placed in the lateral decubitus position with the affected side up and a Dutchman's roll or pillow under the iliac crest. Positioned at the edge of the table, the patient's inferior leg is flexed with the foot at the table's edge. The patient grasps the headpiece of the table with the superior hand, allowing the superior leg to drop off the back of the table.The therapist stands behind the patient, providing support to prevent posterior pelvic rotation with their thigh behind the pelvis. The cephalad hand grasps the top of the iliac crest and applies a caudad force, while the caudad hand gently guides the affected leg without generating force.The patient "hikes" the hip against the resistance from the therapist's cephalad hand, creating an isometric contraction for 5-10 seconds. The patient then relaxes, followed by a rapid stretch held for 10 seconds until the next barrier is reached. This procedure is repeated 3-5 times.
  Arms: PFS Group
Other: Reciprocal Inhibition — The patient is placed in the lateral decubitus position with the affected side up and a Dutchman's roll or pillow under the iliac crest. Positioned at the edge of the table, the patient's inferior leg is flexed with the foot at the table's edge. The patient grasps the headpiece of the table with the superior hand, allowing the superior leg to drop off the back of the table.The therapist stands behind the patient, providing support to prevent posterior pelvic rotation with their thigh behind the pelvis. The cephalad hand grasps the top of the iliac crest and applies a caudad force, while the caudad hand gently guides the affected leg without generating force.The patient "hikes" the hip against the resistance from the therapist's cephalad hand, creating an isometric contraction for 5-10 seconds. The patient then relaxes, followed by a rapid stretch held for 10 seconds until the next barrier is reached. This procedure is repeated 3-5 times.
  Arms: RI Group
Other: Conventional Physical Therapy — A comprehensive therapeutic regimen that includes a 10-minute session of hot pack therapy specifically targeted at the low back region. In addition to this, participants will receive trigger point release therapy to alleviate muscle tension.The treatment plan also incorporates a tailored exercise protocol designed to enhance back health and strength. This protocol includes:
  1. Back isometric exercises
  2. Bridging exercises
  3. Cat and camel stretches
  4. Prone press-ups
  5. Abductor strengthening exercises

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the effects Post facilitation stretch versus reciprocal inhibition on pain, lumbar range of motion, apparent leg length discrepancy and lumbar lordotic angle in Quadratus Lumborum Syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to determine the difference between Post facilitation, stretch versus reciprocal inhibition on pain, lumbar range of motion, apparent leg length discrepancy and lumber lordotic angle in Quadratus Lumborum Syndrome.

The individual of Age 18-35 years among both genders, who experiences pain of 3 ≤ on NPRS from at least 3 months and whose pain decreases on supine lying; along with any two of the following findings positive of quadratus lumborum on physical examination i.e., Taut bands, Local tenderness, Patient's pain recognition, Pain referral to greater trochanter, Local twitch response & Jump sign will be recruited in the study as patients of Quadratus lumborum syndrome.

Pain levels will be assessed using the Numeric Pain Rating Scale (NPRS). Inclinometer will be used for measuring lumber ranges. To assess apparent leg length discrepancy measuring tape will be used. The lumbar lordotic angle will be measured using 60 cm flexible ruler. Participants of interest would be approached and explained about the research. Informed written consent will be taken. It is a non-blinded study and randomization will be done through sealed envelope. Both groups will receive conventional intervention. Additionally, Group A will receive quadratus lumborum post facilitation stretches while Group B will receive Reciprocal inhibition. Baseline and post intervention scores would be recorded for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Both genders
* Having pain of ≤ 8 on NPRS from at least 3 months
* Pain decreases on supine lying
* Any two of the following findings positive of unilateral quadratus lumborum on physical examination:

  1. Taut bands
  2. Local tenderness
  3. Patient's pain recognition
  4. Pain referral to greater trochanter
  5. Local twitch response

Exclusion criteria:

* Painful isometric muscle testing of hip flexors, abductors, adductors, and extensors
* Previous surgery of lower limb
* Centralization/peripheralization
* Lower back trauma
* Positive SLR
* Radiculopathy
* Fracture/surgery of pelvic and/or hip region
* Diagnosed fibromyalgia or other rheumatic diseases.
* Lactating women
* Intrauterine device
* Pregnant women
* Use of psychiatric medications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Pain is assessed by using numeric main rating scale comparing pre and post pain intensity. This is 11- point numeric scale ranges from '0' representing one pain extreme (e.g., "no pain") to '10' representing the other pain extreme
Lumbar Range of Motion (ROM) | 2 weeks
  It will measured using inclinometer
Leg Length Discrepancy (LLD) | 2 weeks
  Measure the distance between the anterior superior iliac spine (ASIS) and the medial malleolus.This method, referred to as the "direct" clinical method for measuring LLD, provides the apparent leg length discrepancy.
Lumbar Lordotic Angle | 2 weeks
  It will be measured using Flexible Ruler

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan